CLINICAL TRIAL: NCT06456463
Title: A Phase II Multicenter Open-label Trial of Tagraxofusp (Tag) in Combination With Venetoclax and Azacitidine (Ven/Aza) in Adults With Previously Untreated CD123+ Acute Myeloid Leukemia (AML) Who Are Ineligible for Intensive Chemotherapy
Brief Title: A Study of Tagraxofusp in Combination With Venetoclax and Azacitidine in Adults With Untreated CD123+ Acute Myeloid Leukemia Who Cannot Undergo Intensive Chemotherapy
Acronym: TRILLIUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STML-401-0423; U1111-1290-9087 (Other: UTN); 2024-514660-48 (Other: EU CT Number)
Record Dates: First submitted 2024-05-31; First posted 2024-06-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: CD123+; Tagraxofusp; Venetoclax; Azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tagraxofusp; Product Labeling; venetoclax; Azacitidine

STUDY DESIGN:
Intervention Model Description: Part 1 (randomized) will evaluate 2 dose levels of tagraxofusp in parallel. The decision to proceed to Part 2 (non-randomized) will be based upon review of cumulative data from Part 1.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 - Tagraxofusp (9 μg/kg/day) (Experimental): Participants will receive tagraxofusp in combination with venetoclax and azacitidine.
  Interventions: Drug: Tagraxofusp; Drug: Venetoclax; Drug: Azacitidine
- Part 1 - Tagraxofusp (12 μg/kg/day) (Experimental): Participants will receive tagraxofusp in combination with venetoclax and azacitidine.
  Interventions: Drug: Tagraxofusp; Drug: Venetoclax; Drug: Azacitidine
- Part 2 - Tagraxofusp (Selected Dose) and TP53 Wild Type (Experimental): Participants (TP53 wild type) will receive tagraxofusp in combination with venetoclax and azacitidine.
  Interventions: Drug: Tagraxofusp; Drug: Venetoclax; Drug: Azacitidine
- Part 2 - Tagraxofusp (Selected Dose) and TP53 Mutated (Experimental): Participants (TP53 mutated) will receive tagraxofusp in combination with venetoclax and azacitidine.
  Interventions: Drug: Tagraxofusp; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Tagraxofusp — Tagraxofusp will be administered by intravenous infusion for 3 consecutive days during each 28-day cycle.
  Other Names: Tag; Elzonris
Drug: Venetoclax — Venetoclax will be administered as an oral tablet (400 milligrams [mg]) daily, with ramp up in Cycle 1, and should be continued at target dose (400 mg) for the remainder of Cycle 1 and subsequent cycles of 28 days each.
  Other Names: Ven; Venclexta
Drug: Azacitidine — Azacitidine will be administered subcutaneously or by intravenous infusion (75 milligrams/square meter) over 7 days of each 28-day cycle, per institutional guidelines/physician choice.
  Other Names: Aza; Vidaza

SUMMARY:
This study will be divided into 2 parts (Part 1 and Part 2). Part 1 will evaluate 2 doses of tagraxofusp (9 and 12 micrograms/kilogram/day [μg/kg/day]), used in combination with venetoclax and azacitidine, to determine the dose for Part 2. This determined dose, in combination with venetoclax and azacitidine, will then be further evaluated in Part 2 in 2 cohorts (TP53 mutated and TP53 wild type). Both parts will be conducted in participants with previously untreated CD123+ AML who are ineligible for intensive chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Previously untreated with histological confirmation of AML by World Health Organization 2022 criteria and are ineligible for treatment with a standard cytarabine and anthracycline induction regimen due to age, or comorbidity.
* Participant has any level of CD123 expression on blasts.
* Participants must be considered ineligible for intensive chemotherapy, defined by the following:

  * ≥75 years of age; or
  * ≥18 to 74 years of age with at least 1 of the following:

    * Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3.
    * Diffusing capacity of the lung for carbon monoxide of ≤65% or forced expiratory volume in 1 second ≤65%.
    * Baseline creatinine clearance ≥30 to <45 milliliters/minute calculated by the Cockcroft Gault formula or measured by 24-hour urine collection.
    * Hepatic disorder with total bilirubin >1.5 x upper limit of normal.
    * Any other condition for which the physician judges the participant to be unsuitable for intensive chemotherapy.
* ECOG performance status:

  * 0 to 2 for participants ≥75 years of age, or
  * 0 to 3 for participants ≥18 to 74 years of age.

Key Exclusion Criteria:

* Participant has received prior therapy for AML.
* Participant is willing and able to receive standard induction therapy.
* Participant has received treatment for an antecedent hematologic disease with a hypomethylating agent, venetoclax, tagraxofusp, purine analogue, cytarabine, intensive chemotherapy, SCT, chimeric antigen receptor-T therapy, or other experimental therapies.
* Participant has AML with central nervous system involvement.

Note: Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-02-09 (Estimated); Study Completion 2030-02-11 (Estimated)

PRIMARY OUTCOMES:
Part 1: Determination of Part 2 Selected Dose of Tagraxofusp When Administered in Combination with Venetoclax and Azacitidine | Cycles 1-4 (up to 112 days; 28 days/cycle)
Part 2: Number of Participants Achieving a Best Overall Response (BOR) of Complete Remission (CR) | Cycles 1-4 (up to 112 days; 28 days/cycle)

SECONDARY OUTCOMES:
Parts 1 and 2: Number of Participants Achieving a BOR of CR | Cycles 1-6 (up to 168 days; 28 days/cycle)
Parts 1 and 2: Time to First CR | Cycles 1-6 (up to 168 days; 28 days/cycle)
  The time to first CR will be defined as the time from randomization (Cycle 1, Day 1) to the date of first documented CR.
Parts 1 and 2: Duration of Response | Cycles 1-6 (up to 168 days; 28 days/cycle)
Parts 1 and 2: Number of Participants Achieving a BOR of CR, CR with Incomplete Hematologic Recovery (CRi), or CR with Partial Hematologic Recovery (CRh) | Cycles 1-4 (up to 112 days; 28 days/cycle)
Parts 1 and 2: Time to First Composite CR | Cycles 1-4 (up to 112 days; 28 days/cycle)
  The time to first composite CR will be defined as the time from randomization (Cycle 1, Day 1) to the date of first documented CR, CRi, or CRh.
Parts 1 and 2: Number of Participants Achieving a BOR of CR or CRi | Cycles 1-6 (up to 168 days; 28 days/cycle)
Parts 1 and 2: Time to first CR/CRi | Cycles 1-6 (up to 168 days; 28 days/cycle)
  The time to first CR/CRi will be defined as the time from randomization (Cycle 1, Day 1) to the date of first documented CR or CRi.
Parts 1 and 2: Event-free Survival (EFS) | Up to approximately 6 years
  EFS will be defined as the time from the date of randomization (Cycle 1, Day 1) until the date of treatment failure, hematologic relapse after CR/CRi/CRh, or death from any cause, whichever occurs first.
Parts 1 and 2: CR with Minimal Residual Disease (MRD) Negative | Cycles 1-6 (up to 168 days; 28 days/cycle)
  Defined as the number of participants with a presence of marrow MRD of less than 0.01% at the time of CR.
Parts 1 and 2: Number of Participants Who Bridged to Stem Cell Transplant (SCT) Through Study Treatment | Up to approximately 6 years
Part 1: Plasma Concentration of Free Tagraxofusp, Venetoclax, and Azacitidine | Predose, up to 8 hours post dose (Days 4, 5, 6, 7, 14; Cycles 1-4; 28 days/cycle)
Part 2: Plasma Concentration of Free Tagraxofusp and Venetoclax | Predose, up to 8 hours post dose (Days 4, 5, 6, 7, 14; Cycles 1-4; 28 days/cycle)
Parts 1 and 2: Number of Participants With Serum Anti-drug Antibodies for Tagraxofusp, Venetoclax, and Azacitidine | Day 4 of each cycle (each cycle is 28 days) up to the end of study (approximately 6 years)
Parts 1 and 2: Exposure-response of Free Tagraxofusp When Administered in Combination with Venetoclax and Azacitidine | Up to approximately 6 years
  The exposure-response relationship will be assessed utilizing the CR rate/composite CR rate and the number of participants experiencing adverse events of interest. This model-based analysis will be conducted to compare the exposure and response of free tagraxofusp, venetoclax, and azacitidine with venetoclax and azacitidine. Results will be reported as percent probability, wherein changes in the percent probability would indicate corresponding changes in the response rates with changes in exposure.
Parts 1 and 2: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to approximately 6 years
Parts 1 and 2: Overall Survival | Up to approximately 6 years
Parts 1 and 2: Maximum Plasma Concentration (Cmax) of Tagraxofusp and Venetoclax | Predose, up to 8 hours post dose (Days 4, 5, 6, 7, 14; Cycles 1-4; 28 days/cycle)
Parts 1 and 2: Time to Reach Cmax (Tmax) of Tagraxofusp and Venetoclax | Predose, up to 8 hours post dose (Days 4, 5, 6, 7, 14; Cycles 1-4; 28 days/cycle)
Parts 1 and 2: Area Under the Concentration-time Curve (AUC) of Tagraxofusp and Venetoclax | Predose, up to 8 hours post dose (Days 4, 5, 6, 7, 14; Cycles 1-4; 28 days/cycle)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (25):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford Health Care, Stanford, California
  - University of Miami, Miami, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System Brigitte Harris Cancer Pavillion, Detroit, Michigan
  - Washington University - Siteman Cancer Center, St Louis, Missouri
  - John Theurer Cancer Center - Hackensack Meridian Health, Hackensack, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Derrick L Davis Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Sydney Kimmel (Thomas Jefferson University), Philadelphia, Pennsylvania
  - Sarah Cannon, the Cancer Institute of HCA Healthcare, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor Scott & White Health, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincents Hospital, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Perth Hospital, Perth, Western Australia